CLINICAL TRIAL: NCT02105753
Title: Treatment of Axillary Hyperhidrosis With a 1210nm Diode Laser
Brief Title: Tx Axillary Hyperhidrosis 1210nm Diode Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Candela Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2012.0010
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2014-09

CONDITIONS: Axillary Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1210nm axillary laser treatments (Experimental): two laser treatments right axilla and one treatment left axilla
  Interventions: Device: 1210nm Diode Laser treatments
- 1210nm laser treatments to the axilla (Experimental): two laser treatments left axilla and one treatment right axilla
  Interventions: Device: 1210nm Diode Laser treatments

INTERVENTIONS:
Device: 1210nm Diode Laser treatments

SUMMARY:
Primary axillary hyperhidrosis is a common idiopathic disorder of the eccrine sweat glands that interferes with daily activities and causes significant social distress. This pilot study is designed to evaluate the efficacy and histologic effects of the 1210nm diode laser for the treatment of axillary hyperhidrosis. Initial results may inform the design of an anticipated larger prospective controlled trial. Study participants will receive one laser treatment to one randomly-assigned axilla using the 1210 nm diode laser, and two treatments to the opposite axilla. Changes in sweating will be measured both by quantitative gravimetric analysis of sweat production and by expert panel evaluation of photographs of the starch-iodine test performed on each axilla. Participants will also be asked to subjectively classify the severity of their axillary sweating. These measures will be performed at pretreatment and at one, three, and six months following treatment. Biopsies of both axillae will be done before and two weeks after treatment to assess histologic changes to the eccrine gland and surrounding structures. Treatment of axillary hyperhidrosis with the 1210nm diode laser is a novel approach based on the unique absorption characteristics of this wavelength. We hypothesize that selective heating of lipids at the appropriate tissue level will impact adjacent eccrine glands typically seated at the dermo-hypodermal junction, leading to subjective and/or objective decreases in eccrine secretions. This type of treatment may offer an effective, non-invasive and safe alternative to current treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years old, and no older than age 64.
2. Subjects must have localized hyperhidrosis only (axillae +/- palms of the hands, soles of the feet, face and other localized areas) without evidence of generalized hyperhidrosis.
3. Subjects must be fully informed and read and sign the informed consent.
4. Subjects must be willing and able to comply with all follow-up requirements.
5. Subjects must be willing to allow two biopsies of each axilla.

Exclusion Criteria:

1. Subjects must not be younger than age 18 years or older than age 64
2. Subjects must not have had previous axillary laser hair reduction nor plan to have laser hair reduction while in the study.
3. Subjects must not have had previous surgical treatment of the axillae such as axillary gland excision, liposuction, sympathectomy, or subcutaneous curettage and must be willing to avoid such therapies while in the study.
4. Subjects must not have received axillary injections of botulinum toxin nine months prior to treatment and must be willing to avoid such therapies while in the study.
5. Subjects must avoid use of depilatories to either axilla during the duration of the study
6. Subjects must not have used aluminum chloride within 1 week or had iontophoresis treatment to the axillae one month prior to treatment
7. Subjects must not have a history of systemic disease leading to excess sweating including hyperthyroidism and diabetes mellitus
8. Subjects must not have active local or systemic infection.
9. Subjects must not be immunocompromised.
10. Subjects must not be pregnant or nursing. Pregnancy test will be offered initially and before each treatment if subject is not sure of status.
11. Active duty military subjects who will be deploying within 7 months after accessioned into the study will be excluded
12. Subjects who refuse to sign the informed consent document and/or refuse to comply with all follow-up requirements will be excluded
13. Subjects must sweat a minimum of 100mg per axillae for men and 50mg per axillae for women

    -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
subjective global assessment questionnaire | 7 months
  To evaluate the impact of 1210nm diode laser pulses on sweat output and eccrine gland histology in subjects with axillary hyperhidrosis. Changes in sweat production from a single and double treatment using treatment parameters designed to deliver heat to the dermo-hypodermal junction will be measured. Subjective assessment of outcome will also be measured. The objective and subjective measurement instruments are detailed in the methods section below.Prior to any treatment, baseline level of sweat production will be evaluated with three instruments: A subjective global assessment questionnaire, gravimetric analysis, and the modified starch-iodine test.
gravimetric analysis | 7 months
  To evaluate the impact of 1210nm diode laser pulses on sweat output and eccrine gland histology in subjects with axillary hyperhidrosis. Changes in sweat production from a single and double treatment using treatment parameters designed to deliver heat to the dermo-hypodermal junction will be measured. Subjective assessment of outcome will also be measured. The objective and subjective measurement instruments are detailed in the methods section below.Prior to any treatment, baseline level of sweat production will be evaluated with three instruments: A subjective global assessment questionnaire, gravimetric analysis, and the modified starch-iodine test.
modified starch-iodine test | 7 months
  To evaluate the impact of 1210nm diode laser pulses on sweat output and eccrine gland histology in subjects with axillary hyperhidrosis. Changes in sweat production from a single and double treatment using treatment parameters designed to deliver heat to the dermo-hypodermal junction will be measured. Subjective assessment of outcome will also be measured. The objective and subjective measurement instruments are detailed in the methods section below.Prior to any treatment, baseline level of sweat production will be evaluated with three instruments: A subjective global assessment questionnaire, gravimetric analysis, and the modified starch-iodine test.

CONTACTS AND LOCATIONS:
Overall Officials: John P. Trafeli, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- NMCSD, San Diego, California, United States